CLINICAL TRIAL: NCT03787407
Title: The Effect of Neurofeedback-assisted Mindfulness Training on Stress Reduction in Employees With Emotional Labor
Brief Title: The Effect of Neurofeedback-assisted Mindfulness Training in Employees With Emotional Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ministry of Trade, Industry & Energy, Republic of Korea (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: B-1807/483-303
Record Dates: First submitted 2018-12-23; First posted 2018-12-26 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2018-12

CONDITIONS: Stress, Psychological
Keywords: resilience; emotional labor; mindfulness; neurofeedback
MeSH Terms: conditions — Stress, Psychological | interventions — Meditation

STUDY DESIGN:
Intervention Model Description: Healthy individuals recruited through advertisement
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness training with neurofeedback (Experimental): mindfulness training with neurofeedback using mobile application instruction and review of the application will be provided
  Interventions: Behavioral: stress management and meditation
- Mindfulness training (Active Comparator): mindfulness training using mobile application instruction and review of the application will be provided
  Interventions: Behavioral: stress management and meditation
- Self-care (No Intervention)

INTERVENTIONS:
Behavioral: stress management and meditation — mindfulness training using mobile application
  Arms: Mindfulness training; Mindfulness training with neurofeedback

SUMMARY:
The purpose of this study is to verify the effect of neurofeedback-assisted mindfulness training for workers. Subjects who can participate in the screening are assigned to one neurofeedback-assisted mindfulness training group, mindfulness only training group, and self-treatment group. The neurofeedback-assisted mindfulness group and the mindfulness group meet with psychologist and have education for the mindfulness training with or without neurofeedback respectively, a total of 4 times, once a week. On the other hand, the self-treatment group provides self-education by providing the stress education kit.

DETAILED DESCRIPTION:
After screening, Pre-evaluation is conducted on the subjects who agreed to participate in the study. Pre-assessment includes questionnaires related to stress, emotional labor, resilience, sleep, etc., and includes stress-related physiological measures using HRV, 2 lead EEG. After the pre-evaluation, the neurofeedback-assisted mindfulness and mindfulness training group will have education sessions with a psychologist for 30 minutes at a time, once a week, for a total of 4 sessions (one month for a period). The education includes the instruction of the application including mindfulness training, with or without neurofeedback, and the review for the accomplishment of the training. Participants should follow the instruction and the training schedule which is arranged in advance. On the other hand, for a self-care control, the education sessions are not provided and self-learning materials are provided once a week. The purpose of the study is to find the effectiveness of mindfulness training on reduction of stress and severity of emotional labor. Especially, mindfulness training group with neurofeedback might be expected to show the highest improvement in various clinical scales and biomarkers including EEG and HRV.

ELIGIBILITY:
Inclusion Criteria:

* Workers over the age of 19 and under 65
* In the Perceived Stress Scale 14 points or more
* If you are currently taking medication due to psychiatric illnesses such as depression, anxiety disorder, insomnia, etc., the dose must be stabilized for last 6 months, is expected to have no change in drug dose during the clinical trial
* If you understand the protocol and voluntarily agree to participate
* If you have an Android phone

Exclusion Criteria:

* Age under 19, adult over 65
* If you have dementia, intellectual disability, or other cognitive impairment
* If you have convulsive disorder, stroke, or other neurological disorder
* If you have psychosis such as schizophrenia or bipolar disorder or you have a history
* If you have a disease that can affect the reliability of HRV test, such as heart disease or lung disease.
* Has received non-pharmacological psychiatric or counseling treatment within the current or last 6 months.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline Perceived Stress Scale (PSS) score at 4, 8 weeks | Baseline and after 4, 8 weeks later
  The full name: Perceived Stress Scale - 10 item form 14-item scale developed by Cohen et al. (1983) that emphasizes subjective perception of stress. Measures the degree of perceived unforeseeable, uncontrollable, and overwhelming experience of stress in the past month. Although the 14-item PSS tend to exhibit good reliability, four of the items tend to perform poorly when evaluated using exploratory factor analysis (Cohen et al., 1988). As a result, the PSS is commonly implemented using the 10-item form. The questions are rated on 5-point Likert scale; 0 (never), 1 (almost never), 2 (sometimes), 3 (fairly often), 4 (very often). Higher scores represent worse outcomes. The scores of each scale sum into the total score. Thus the total score ranges from 0 to 40.

SECONDARY OUTCOMES:
Change from baseline Korean Emotional Labor Assessment Tool score | Baseline and after 4, 8 weeks later
  The total of 26 items were Emotional expression and control 5 items, organizational monitoring and management system 4 items, forced customer response 4 items, emotional damage 6 items, organizational protection system 7 items, and organizational protection system is reverse coding and summed up. 4 point Likert scale (1 = not at all, 5 = very much), and the possible total score ranges from 26 to 130 points. The higher the score, the more emotional labor means.
Change from baseline Korean abbreviation of Occupational Stress Scale (KOSS) score | Baseline and after 4, 8 weeks later
  total of 24 items were used, and each item was not at all (from 1 point) to very much (5 points). The higher the score, the more the job stress means. Job demand, Insufficient job control, job insecurity, interpersonal conflict, Organizational system, Lack of reward and Occupational climate.
Change from baseline Patient Health Questionnaire 9 (PHQ-9) score | Baseline and after 4, 8 weeks later
  The total score is 0 to 27, and the higher the total score, the more severe the depressive symptoms. Cutpoints of 5, 10, 15 and 20 represent the thresholds for mild, moderate, moderate severe, and severe depression, respectively.
Change from baseline Brief resilience scale (BRS) score | Baseline and after 4, 8 weeks later
  It is composed of 6 questions and is evaluated on the 5-point scale (1: not at all, 5: very much)
Change from baseline Athens Insomnia Scale (AIS) score | Baseline and after 4, 8 weeks later
  total score of 6 points was used as a breakpoint, this Using the quality index of Pittsburgh Sleep, which is widely used to evaluate the quality of sleep
Korean Mindful Attention Awareness Scale; K-MAAS | Baseline and after 4, 8 weeks later
  Modified from the Mindful Attention Awareness Scale, developed by Brown and Ryan (2003). 15-item scale designed to assess a core characteristic of dispositional mindfulness, namely, open or receptive awareness of and attention to what is taking place in the present.
Stroop test | Baseline and after 4, 8 weeks later
  assess the ability to inhibit cognitive interference that occurs when the processing of a specific stimulus feature impedes the simultaneous processing of a second stimulus attribute
Heart Rate Variability (HRV) | Baseline and after 4, 8 weeks later
  HRV is recorded with a device (neuroNicle FX2, Laxtha) which include EEG and HRV recording system. HRV is calculated from pulse rate signal recorded at earlobe.
Quantitative electroencephalography (QEEG) | Baseline and after 4, 8 weeks later
  EEG is recorded with a device (neuroNicle FX2, Laxtha) which include EEG and HRV recording system. EEG signal is acquired at the prefrontal area, two channels (FP1, FP2) on forehead.
  Power spectrum analysis of the EEG data will be performed using Fourier analysis. And absolute power, relative power, of each frequency band, symmetry are included.

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Hyun Kim, MD, Ph.D, Principal Investigator — Seoul National Univerysity Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Min B, Park H, Kim JI, Lee S, Back S, Lee E, Oh S, Yun JY, Kim BN, Kim Y, Hwang J, Lee S, Kim JH. The Effectiveness of a Neurofeedback-Assisted Mindfulness Training Program Using a Mobile App on Stress Reduction in Employees: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2023 Oct 3;11:e42851. doi: 10.2196/42851. PMID 37788060